CLINICAL TRIAL: NCT06593171
Title: Decreasing the Stigma of Mental Illness Among Health Science Students Through a Mentoring Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Matías E. Rodríguez-Rivas, Principal Investigator, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 815
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Social Stigma
MeSH Terms: conditions — Social Stigma | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): No intervention group
  Interventions: Behavioral: Control (placebo) group
- Experimental group (Experimental): Intervention group. In detail, the intervention has a total of 3 participatory sessions via videoconference, with an average duration of 90 minutes per session, with a maximum number of 3 to 4 students per mentor. Each session is accompanied by a reflective log of the activities and observations made by the students of an evaluated nature, as well as reading prior to session n°1 and n°2. In addition, the anonymous evaluation of the level of stigma before and after the implementation, both in the group of students and mentors, is included, as well as a follow-up of the measurements regarding these evaluations.
  At the professional level, a 6-hour pedagogical intervention focused on stigma reduction for the training of health students towards people with psychiatric illnesses will be provided to all health professionals involved, with a certificate of participation delivered at the end of the sessions.
  The sessions must have minimum material implements such as an equipped classroom, proj
  Interventions: Behavioral: Mentoring program

INTERVENTIONS:
Behavioral: Mentoring program — This three-session mentoring program is based on experiential learning and has been validated and adapted to our country. The mentors, professionals with lived experience in mental health, will provide knowledge and experiences to the students through direct contact sessions in the classroom, focusing especially on the processes of recovery and self-determination.
  Arms: Experimental group
Behavioral: Control (placebo) group — This group will not receive any intervention. However, they will be invited to participate in stigma education after the study is completed.
  Arms: Control group

SUMMARY:
Stigma towards people with mental health problems is a serious public health problem that limits access to treatment and social participation, in addition to being considered the main barrier to inclusion and quality of health care. This stigma also affects students and health professionals, impacting the quality of care and help seeking in mental health. In this context, it is necessary to develop innovative and effective interventions among university students to reduce this stigma and promote an inclusive and recovery-based approach.

The aim of the present research project is to analyze the effect of a mentoring program on levels of stigma and mental health help-seeking intention in psychology and nursing students. This three-session mentoring program is based on experiential learning and has been validated and adapted to our country. The mentors, professionals with lived experience in mental health, will provide knowledge and experiences to the students through direct contact sessions in the classroom, focusing especially on the processes of recovery and self-determination.

Research question: What is the effect of a mentoring program on levels of stigma and mental health help-seeking intention in health care students?

Within the dependent variables of the study are the measurement of levels of stigma and mental health help-seeking intention in students. The independent variables will be the type of group (experimental and control), age, gender and career.

Methodology: Quantitative study, including the participation of health students in the experimental and control groups. The sample size was determined using the G*Power software. After approval by the institutional ethics committee and signature of the informed consent of the participants, the mentoring program will be implemented in the classroom. For this purpose, the levels of stigma and intention to seek mental health help in both groups will be measured using nationally and internationally validated instruments, before, after and at 4 weeks. Data analysis will be performed using a mixed ANOVA model to compare pre- and post-intervention outcomes between the two groups.

The present study will provide valuable evidence on the effectiveness of mentoring-based interventions in reducing stigma in health care students, a key group in the future provision of care for people with mental health problems. The results will also lay the groundwork for larger-scale studies to assess the impact of the intervention in other groups and settings, with the potential to significantly improve the quality of care and well-being of patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* University students from health careers
* Sign the informed consent form.

Exclusion Criteria:

* Be under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Attribution Questionnaire (AQ-27) | At the time of recruitment, immediately after the end of the study and the 4-week follow-up.
  This 27-item, 9-factor instrument has been widely used to measure levels of stigma towards people with mental health problems in the general population and university students nationally and globally. It presents a vignette of a case of a person diagnosed with schizophrenia, where various stereotypes, prejudices and behaviors around him are assessed and measured (anger, pity, dangerousness, fear, avoidance, guilt, segregation and coercion). The instrument uses a 9-point Likert-type response scale, where higher scores represent higher levels of stigma. Specifically, its Spanish version has demonstrated adequate psychometric properties for use in a university population (Saavedra et al., 2021).
Mental Help Seeking Intention Scale (MHSIS) | At the time of recruitment, immediately after the end of the study and the 4-week follow-up.
  A 3-item instrument designed to measure respondents' intention to seek help from a mental health professional if one were to have a mental health problem (Hamer & Spiker, 2018). The response scale is a 7-point Likert-type, where a higher score indicates a greater intention to seek help. This instrument has been shown to possess psychometric properties suitable for use with college students, in addition to possessing evidence of predictive validity (Hamer & Spiker, 2018).